CLINICAL TRIAL: NCT01769768
Title: A Phase Ib, Multi-center, Two Parallel Group, Open-label, Drug-drug Interaction Study to Assess the Effect of LDE225 on the Pharmacokinetics of Bupropion and Warfarin in Patients With Advanced Solid Tumors
Brief Title: Phase I Study to Evaluate the Effect of LDE225 on the Pharmacokinetics of Bupropion and Warfarin in Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDE225A2112
Record Dates: First submitted 2013-01-15; First posted 2013-01-17 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2017-02

CONDITIONS: Advanced Solid Tumor
Keywords: Adults, Hh (Hedgehog) pathway inhibitor, LDE225, Warfarin, Bupropion, advanced solid tumor, drug-drug interaction, pharmacokinetic
MeSH Terms: interventions — sonidegib; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- LDE225+Warfarin (Experimental): At least 15 evaluable patients with advanced solid tumors will be enrolled into the study into the warfarin group.
  Interventions: Drug: LDE225; Drug: Wafarin
- LDE225+Bupropion (Experimental): At least 15 evaluable patients with advanced solid tumors will be enrolled into the study into the Bupropion group
  Interventions: Drug: LDE225; Drug: Bupropion

INTERVENTIONS:
Drug: LDE225 — LDE225 800 mg once daily dosing will begin on Cycle 1 Day 1 of a 28-day cycle.Treatment with LDE225 for both groups will continue until the patient experiences unacceptable toxicity that precludes further treatment, disease progression, withdrawal of consent and/or at the discretion of the investigator.
Drug: Wafarin — 15 mg single dose of warfarin (oral tablet) will be given to patients.
  Arms: LDE225+Warfarin
Drug: Bupropion — 75 mg single dose of bupropion(oral tablet, from an immediate release formulation) will be given to patients
  Arms: LDE225+Bupropion

SUMMARY:
This is a multi center, open-label study to evaluate the drug-drug interaction of LDE225 on the PK of bupropion and warfarin patients with advanced solid tumors. Subjects will receive 800mg daily of LDE225 and two separate doses of either bupropion or warfarin.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Patients with cytopathologically or histopathologically confirmed diagnosis of an advanced solid tumor which has progressed despite standard therapy, or for which no standard therapy exists or patients with locally advanced or metastatic basal cell carcinoma who are not amendable or eligible for standard therapy.
* Protocol-defined renal , liver and bone marrow function

Exclusion Criteria:

* CNS (Central Nervous System) tumors as well as history of brain metastases
* Systemic anticancer treatment (including biologic therapy/antibodies) within 2 weeks before first dose of study treatment (6 weeks for nitrosourea, mitomycin, and monoclonal antibodies).
* Radiation therapy within 4 weeks before first dose
* Investigational agents within 4 weeks before start of study therapy
* Patients with known allergy/hypersensitivity to warfarin or bupropion and/or related compounds
* Patients with a history of/or active bleeding disorders
* Patients receiving treatment with vitamin K, Coumadin or other agents containing warfarin and heparin. Heparin flush to maintain patency of a central venous access device is allowed.
* Patients receiving treatment with bupropion.
* Patients who have neuromuscular disorders that are associated with elevated CK (Creatine phosphokinase) (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy).
* Known diagnosis of human immunodeficiency virus (HIV), Hepatitis B or C (testing is not mandatory for study entry)
* Patients currently receiving systemic corticosteroids

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2013-04; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) parameter AUClast for S- and R-warfarin | 7 days
  Pharmacokinetics of warfarin : Maximum observed plasma concentration after drug administration
PK parameter AUClast for bupropion | 7 days
  Pharmacokinetics bupropion : Maximum observed plasma concentration after drug administration
PK parameter AUCinf for bupropion | 7 days
  Pharmacokinetics of bupropion : Maximum observed plasma concentration after drug administration
PK parameter AUCinf for S- and R-warfarin | 7 days
  Pharmacokinetics of warfarin and bupropion : Maximum observed plasma concentration after drug administration
PK parameter Cmax for S- and R-warfarin | 7 days
  Pharmacokinetics of warfarin : Maximum observed plasma concentration after drug administration
PK parameters Cmax for bupropion | 7 days
  Pharmacokinetics of Bupropion : Maximum observed plasma concentration after drug administration

SECONDARY OUTCOMES:
effects of LDE225 on the pharmacodynamic activity of warfarin | 7 days
  INR parameter (International Normalized Ratio) will be assessed to evaluate the pharmacodynamic effect of warfarin.
safety of LDE225 when administered alone and concomitantly with either bupropion or warfarin | 28 days cycles
  safety laboratory parameters, adverse event reports, changes in vital signs, changes in physical examination parameters
evaluate the preliminary evidence of anti-tumor activity of LDE225 in patients with advanced solid tumors | every other cycle
  CT or MRI imaging parameters to determine the objective response rate according to RECIST 1.1 (Response Evaluation Criteria In Solid Tumors)
assess the effect of LDE225 treatment on cardiac function | screening, cycle 4 and EOT
  ECGs will be performed to determine the effect of LDE on the cardiac function.
effects of LDE225 on the pharmacodynamic activity of warfarin | 7 days
  PT (Prothrombin time) parameter will be assessed to evaluate the pharmacodynamic effect of warfarin.
safety of LDE225 when administered alone and concomitantly with either bupropion or warfarin | 28 days cycles
  safety laboratory parameters
safety of LDE225 when administered alone and concomitantly with either bupropion or warfarin | 28 days cycles
  adverse event reports
safety of LDE225 when administered alone and concomitantly with either bupropion or warfarin | 28 days cycles
  changes in vital signs

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (13):
  - City of Hope National Medical Center Oncology, Duarte, California
  - University of Kansas Medical Center CBYM338B2203, Kansas City, Kansas
  - Massachusetts General Hospital Dana-Farber Cancer Institute, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Dartmouth Hitchcock Medical Center Dartmouth-Hitchcock Med Ctr, Lebanon, New Hampshire
  - Hackensack University Medical Center Dept.of HackensackUniv.MedCtr., Hackensack, New Jersey
  - University of Pennsylvania--Abramson Cancer Center Abramson Cancer Center, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - University of Pittsburgh Cancer Institute UPMC Cancer Pavilion, Pittsburgh, Pennsylvania
  - Medical University of South Carolina Dept.of Neurosciences/MS Ctr., Charleston, South Carolina
  - Cancer Centers of the Carolinas SC, Greenville, South Carolina
  - Utah Health Science Center at San Antonio, San Antonio, Texas
  - University of Utah / Huntsman Cancer Institute, Salt Lake City, Utah

REFERENCES:
- [Derived] Pooler DB, Ness DB, Sarantopoulos J, Squittieri N, Ravichandran S, Britten CD, Amaravadi RK, Vaishampayan U, LoRusso P, Shapiro GI, Olszanski AJ, Perez R, Gutierrez M, O'Rourke MA, Chung V, Lee JJ, Lewis LD. The effect of sonidegib (LDE225) on the pharmacokinetics of bupropion and warfarin in patients with advanced solid tumours. Br J Clin Pharmacol. 2021 Mar;87(3):1291-1302. doi: 10.1111/bcp.14508. Epub 2020 Aug 20. PMID 32736411
- See also: Results for CLDE225A2112 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=16289